CLINICAL TRIAL: NCT03019328
Title: Early Peanut Introduction: Translation to Clinical Practice
Acronym: EPI
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00095833; 1U01AI125290 (NIH)
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Peanut Allergy
Keywords: peanut allergy; food allergens; atopic dermatitis; eczema; infant food allergy testing; skin prick testing; peanut IgE; early peanut introduction; food allergy prevention
MeSH Terms: conditions — Peanut Hypersensitivity; Dermatitis, Atopic; Eczema | interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloods, skin swabs, skin tape strips
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Peanut in diet

SUMMARY:
The recent finding that early introduction of peanut can prevent ~70-90% of peanut allergy is a major step towards prevention of food allergy. However, because that finding was from a clinical trial in a very select population, there are several major questions that must be answered in order to implement these findings into clinical practice without causing more harm than good. These questions include who, if anyone, should be screened prior to early introduction for peanut allergy, how this screening should be done, and what quantity of peanut ingestion is needed to prevent peanut allergy. The goal of this project is to answer these critical questions so that the potential of these recent findings can be realized. To that end, 400 infants at high-risk of peanut allergy will be enrolled. These infants will be given a peanut skin prick test, peanut food challenge and have blood drawn for measurement of peanut IgE, and then will be followed for assessment of peanut consumption and development of peanut allergy until 3 years of age.

DETAILED DESCRIPTION:
400 infants aged 4-11 months from three high risk groups will be enrolled in a prospective observational study. All subjects will have a baseline research clinic visit, where they will be given a peanut skin prick test, peanut food challenge and have blood drawn for measurement of peanut immunoglobulin E (IgE). Based on the baseline oral food challenge, the participants will be advised to begin introducing peanut following the current practice guidelines. Participants will then be followed until 30 months of age with two clinic visits and regular monitoring of peanut consumption.

ELIGIBILITY:
Inclusion Criteria:

* Infants age 4-11 months
* Have at least one of the following criteria:

  1. physician diagnosis of milk, egg or other non-peanut food allergy,
  2. at least moderate eczema as defined by a SCORAD score of at least 25 on present or previous evaluation, OR a rash that required the application of topical creams or ointments containing corticosteroids or calcineurin inhibitors and occurred on at least 7 days on two separate occasions, or is described by the parent or guardian as "a bad rash in joints or creases" or "a bad itchy, dry, oozing or crusted rash".
  3. a first degree relative (parents or siblings) with either a physician diagnosis of IgE mediated peanut allergy OR reported history of symptoms consistent with IgE mediated peanut allergy (onset of symptoms within 2 hours of exposure, AND symptoms of urticaria, angioedema, wheezing, vomiting, or abdominal pain with exposure, AND no subsequent exposure to peanut without symptoms).

Exclusion Criteria:

* History of feeding problems
* History of eosinophilic gastro-intestinal disease
* Significant medical history (aside from eczema, food allergy or history of wheeze)
* History of peanut reactions or tolerance prior to baseline screening

Ages: 4 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants age 4 monhts to 11 months
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Percent of infants with peanut allergy at baseline | Baseline
  Percentage of infants who fail the peanut challenge at the baseline visit

SECONDARY OUTCOMES:
Compare results of peanut skin prick test to peanut challenge outcomes among the high risk infants | baseline
  Results of peanut skin prick tests compared to peanut challenge among the high risk infants
Compare results of anti-peanut IgE testing to peanut challenge outcomes among the high risk infants | baseline
  Results of anti-peanut IgE testing compared to peanut challenge among the high risk infants
Compare results of anti-Ara h2 IgE testing to peanut challenge outcomes among the high risk infants | baseline
  Results of anti-Ara h2 IgE testing compared to peanut challenge among the high risk infants
Percent of infants who develop peanut allergy by age 30 months | 30 months
  Percent of infants at risk who develop peanut allergy during the study window (30 months)
Percent of infants with a skin prick test of 3 mm or more at baseline who develop peanut allergy | 30 months
  Percent of infants with a positive skin prick test who develop peanut allergy during the study window (30 months)
Peanut levels in bedroom dust as measured by home dust collection | 18 months
  Peanut levels will be tested by Elisa in bed dust collected by patients using a DUSTREAM(R) vacuum adaptor.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Keet, MD, Principal Investigator — Johns Hopkins University; Robert Wood, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No